CLINICAL TRIAL: NCT04841330
Title: Prospective Healthy Volunteer Study of the Securis™ Stabilization Device
Status: Completed | Type: Observational
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: MDS-20SECUR001
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Peripheral Intavenous Catheter Stabilization

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Healthy volunteers: A minimum of 100 healthy volunteer participants (14yo and older)
  Interventions: Device: Securis™ Stabilization Device

INTERVENTIONS:
Device: Securis™ Stabilization Device — A trained clinician will apply and remove, and participants will wear the Securis™ Stabilization Device for up to one week (7 days) on their forearm. A shortened catheter will be placed (not inserted) over the Securis™ device in accordance with the product Information for Use (IFU), and an extension set attached to the catheter and secured in place, to simulate clinical use.

SUMMARY:
This study is being conducted to assess the performance of the Securis™ Stabilization Device in simulated clinical use.

DETAILED DESCRIPTION:
This study is designed to collect prospective observational data related to the safety and performance of the Securis™ Stabilization Device in healthy volunteers utilizing a simulated use method. Participants will have an intravenous catheter applied (not inserted) onto their forearm with a Securis™ Stabilization Device applied over it. The site/device will be assessed over a period of 9 days (ideally Days 0-7 in-clinic and Day 8 virtually). The assessments will include the appearance of the site, the appearance of the dressing, and the movement of the catheter tip under the dressing.

ELIGIBILITY:
Inclusion Criteria:

1. ≥14 years of age, regardless of gender, at the time of informed consent
2. Is expected to be available through Day 8 of the study
3. Is expected to understand and follow the study procedures including applicable restrictions in activities (e.g., limited physical exercise, no swimming, no use of lotions/moisturizers, etc.)
4. Provision of signed and dated informed consent form. Note: Consent of a parent of legal guardian will be require for participants <18 years of age; assent will also be required for these participants

Exclusion Criteria:

1. Significant scarring at the device application site
2. Has any skin condition that might affect device adherence or the ability of study staff to perform skin assessments
3. Has any condition or is taking any medication that might cause excessive bruising, bleeding, or skin tearing (e.g., anti-coagulant therapy)
4. Known allergy to study device/components or ancillary devices
5. Will be unable to complete a remote visit via video chat, if required
6. Has any condition which, in the opinion of the Investigator, precludes them from participation in this study.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Potential participants will be recruited from healthy volunteer participant pools identified and/or held by the study site.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Rate of Securis™ Stabilization Device Securement Failure During Simulated Use | From time of placement and up to 8 days after removal
  Device securement failure is defined as any of the following:
  * Loose dressing
  * Soiled under dressing
  * Complete failure (complete removal)
  * Dislodgement of device or catheter
Percentage of Participants with Select Skin Conditions Observed During Securis™ Stabilization Device Use | From placement and up tp to 24 hours after device removal
  Select skin conditions include any of the following:
  * Blister
  * Rash
  * Skin tear
  * Bruising
  * Exudate

SECONDARY OUTCOMES:
Rate of Securis™ Stabilization Device-related Adverse Events | From placement and up to 24 hours after device removal
  Rate of device-related adverse events calculated as the number of participants with adverse events related to the device divided by the total number of evaluable participants.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Casser, MD, Principal Investigator — TKL Research, Inc.
Locations (1):
- TKL Research, Inc, Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided